CLINICAL TRIAL: NCT06281327
Title: A Prospective, One-arm and Open Clinical Study to Assess Efficacy and Safety of Avatrombopag in the Treatment of Pediatric Primary Immune Thrombocytopenia
Brief Title: Avatrombopag in the Treatment of Pediatric Immune Thrombocytopenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Henan Cancer Hospital (Other Government); Tianjin Medical University Second Hospital (Other); Tianjin Children's Hospital (Other); The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2023062
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Immune Thrombocytopenia; Treatment
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — avatrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group: Avatrombopag (Experimental): Sixty subjects will be enrolled with the indicated treatment dose of avatrombopag
  Interventions: Drug: Avatrombopag

INTERVENTIONS:
Drug: Avatrombopag — After enrollment, all subjects receive Avatrombopag treatment. The initial dose of Avatrombopag administration was an oral 10 mg (<30kg) or 20mg (≥30kg) once daily in all participants. ps. For subjects weighing ≥30kg, the dose can be started from 40mg once daily if the platelet count is < 10×10^9/L or if there is severe bleeding or risk of bleeding.
  Complete blood count including platelet count was done once a week. The dose of Avatrombopag was adjusted according to the subject platelet count during the period from week 1 to week 24. If the platelet count was less than 30×10^9/L for 2 weeks, avatrobopag was gradually increased. If the platelet count was greater than 150 x 10^9/L, avatrobopag was gradually reduced. If the platelet count >250×10^9/L, avatrobopag will be stoped until the platelet count <100×10^9/L.

SUMMARY:
To evaluate the safety and efficacy of avatrombopag in the treatment of pediatric primary immune thrombocytopenia in patients who have been treated with eltrombopag before and switched to avatrobopag because of poor efficacy, excessive platelet fluctuation or intolerance, or patient preference, economic reasons, and other reasons.

DETAILED DESCRIPTION:
Immune thrombocytopenia (ITP) is an organ-specific autoimmune disease, which is characterized by decreased platelet count and skin and mucosal bleeding. ITP is a kind of disease with increased platelet destruction and impaired platelet production caused by autoimmunity. Conventional treatment of adult ITP includes first-line glucocorticoid and immunoglobulin therapy, second line TPO and TPO receptor agonist, splenectomy and other immunosuppressive treatments (such as rituximab, vincristine, azathioprine, etc.).

Eltrombopag is currently the only TPO receptor agonist with indications for pediatric immune thrombocytopenia. However, at present, the treatment response of pediatric ITP is not good, and a considerable number of patients need to switched to other TPO receptor agonist, such as avatrombopag, because of poor efficacy, excessive platelet fluctuation or intolerance, or patient preference, economic reasons, and other reasons.

Therefore, the investigators designed this clinical trial to evaluate the efficacy and safety of avatrombopag in the treatment of pediatric immune thrombocytopenia in patients who who have been treated with eltrombopag before and switched to avatrobopag because of different reasons.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-18 years old (including both ends), male and female;
* Diagnosed with primary immune thrombocytopenia (ITP);
* Patients who had previously received eltrombopag treatment and then converted to avatrombopag treatment because of ineffectiveness (platelet count < 30×10^9/L after eltrombopag treatment, or platelet count increased less than 2 times of the basic value, or bleeding) or large platelet fluctuation or due to patient preference, economic reasons and other reasons;
* Cardiac function of the New York Society of Cardiac Function ≤ 2;
* Understand the study procedure and voluntarily sign the informed consent.

Exclusion Criteria:

* Secondary thrombocytopenia caused by various reasons, such as connective tissue disorders, bone marrow hematopoietic failure disease, myelodysplastic syndrome, malignancy, drugs, inherited thrombocytopenia, common variable immune deficiency, lymphoma, etc.;
* Subjects with primary disease of important organs (liver, kidney, heart, etc.), or with immune system diseases;
* Subjects who are known to be allergic to avatrombopag or any of its excipients;
* Subjects who had used rituximab within the last 3 months;
* Subjects who underwent splenectomy within the last 3 months；
* Subjects with a history of abnormal platelet aggregation that may affect the reliability of platelet count measurements；
* Any medical history or condition that the investigator deems unsuitable for participation in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Overall efficacy response after AVA treatment within 12 weeks | 12 weeks
  Overall response rate defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding at the meanwhile within 12 weeks after initial administration in absence of rescue therapy.

SECONDARY OUTCOMES:
Treatment response-1 | 12 weeks
  Number of participants achieving a platelet count ≥ 50×10^9/L at week 1,2,4,6,8,12 in absence of rescue therapy.
Treatment response-2 | 12 weeks
  Number of participants achieving a platelet count ≥ 100×10^9/L at week 1,2,4,6,8,12 in absence of rescue therapy.
Time to Response | 12 weeks
  The time required from the start of treatment to the first time a subject's platelet count was greater than or equal to 30×10^9/L and at least a two-fold increase from the baseline platelet count without bleeding in absence of rescue therapy.
Persistent response | 12 weeks
  Persistent response defined as proportion of subjects with a platelet count ≥ 30 × 10^9/L and at least 2-fold from baseline without bleeding for 4 consecutive weeks or more within 12 weeks after initial administration in absence of rescue therapy.
Emergency treatment | 12 weeks
  The proportion of subjects receiving emergency treatment
Reduction of concomitant drug | 12 weeks
  Percentage of patients with reduced doses of concomitant drugs at baseline
Number of participants with clinically significant bleeding as assessed using the world health organization (WHO) bleeding scale. | 12 weeks
  The WHO Bleeding Scale is a measure of bleeding severity with the following grades: grade 0 = no bleeding, grade 1= petechiae, grade 2= mild blood loss, grade 3 = gross blood loss, and grade 4 = debilitating blood loss.
Number of participants with clinically significant bleeding as assessed using the bleeding scale for pediatric patients with ITP. | 12 weeks
  The bleeding scale for pediatric patients with ITP is a measure of bleeding severity with the following grades: Grade 1 (minor) Minor bleeding, few petechiae (≤100 total) and/or ≤5 small bruises (≤3 cm in diameter), no mucosal bleeding；Grade 2 (mild) Mild bleeding, many petechiae (>100 total) and/or >5 large bruises (>3 cm in diameter), no mucosal bleeding；Grade 3 (moderate) Moderate bleeding, overt mucosal bleeding, troublesome lifestyle；Grade 4 (severe) Severe bleeding, mucosal bleeding leading to decrease in Hb>2 g/dL or suspected internal hemorrhage；
Health-related quality of life survey of subjects(HRQoL)-1 | 12 weeks
  In all participants ,use ITP-PAQ (ITP Patient Assessment Questionnaire) to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-2 | 12 weeks
  In all participants ,use FACIT-F（functional assessment of chronic illness therapy- fatigue）to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-3 | 12 weeks
  In all participants ,use Kids' ITP tool KIT、to assess the HRQoL before and after treatment.
Health-related quality of life survey of subjects(HRQoL)-4 | 12 weeks
  In all participants ,use Pediatric Quality of Life Inventory PedsQL to assess the HRQoL before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Tianjin, China